CLINICAL TRIAL: NCT00645580
Title: Alterations in mRNA and Protein Expression in Human Peripheral Mononuclear Blood Cells (PMC) of Schizophrenia Patients Treated With Fluvoxamine Augmentation of Antipsychotics: Relationship to Clinical Symptoms and Cognitive Function
Brief Title: Genetic Expression in Schizophrenics Treated With SSRI Augmentation: Relationship to Clinical and Cognitive Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sha'ar Menashe Mental Health Center (Other)
Responsible Party: Prof. Henry Silver, Sha'ar Menashe Mental Health Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1-3-08
Record Dates: First submitted 2008-03-23; First posted 2008-03-27 (Estimated); Last update posted 2009-02-19 (Estimated); Status verified 2008-03

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Fluvoxamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: Fluvoxamine

INTERVENTIONS:
Drug: Fluvoxamine — Fluvoxamine 100mg/day PO for 6 weeks.
  Other Names: Favoxil; Luvox; Dumyrox; Fevarin; Faverin

SUMMARY:
In our study we aim to examine the effect of SSRI augmentation on negative symptoms and cognitive function in schizophrenia patients as well as to examine the effect of SSRI augmentation on the RNA and protein products in peripheral mononuclear cells (PMC). Finally, we aim to relate changes in PMC elements to changes in clinical symptoms and cognitive function. Our study hypotheses are that SSRI augmentation of anti-psychotic treatment in schizophrenia patients will improve negative symptoms as well as cognitive symptoms and that this improvement will be related to biochemical changes identifiable in PMC elements.

DETAILED DESCRIPTION:
Clinical studies have shown that adding selective serotonin reuptake inhibitor (SSRI) antidepressants to antipsychotics can improve negative symptoms of schizophrenia in patients unresponsive to antipsychotics alone (Silver and Nassar, 1992; Spina et al., 1994; Goff et al., 1995). However, the effect of SSRI augmentation on cognitive impairments of the illness has not been adequately tested.

The mechanism of SSRI augmentation is not known and is the focus of research interest.

We have recently shown that in animals, combined treatment of SSRI antidepressant and antipsychotic drug resulted in biochemical changes, different from the effects of the individual medications. Changes unique to the combined treatment were found in GABAergic components (GABA-Aβ3 receptor, glutamic acid decarboxylase 67 and PKCβ (Chertkow et al., 2005)) and changes unique to the combined treatment were found in selected areas of rat brain.

Studies of drug mechanisms in humans have utilized blood products and PMC which are readily accessible and may reflect molecular processes in the central nervous system (CNS) of schizophrenic patients (Kronfol and Remick, 2000; Avissar et al., 2001; Ilani et al., 2001; Rothermundt et al., 2001). In a recent study (Chertkow et al., 2007) which examined the gene expression profile of PMC's from antipsychotic-treated patients before the addition of the SSRI fluvoxamine, we found that mRNA expression of chemokine receptors, IL8RA and CCR1, and of RGS7 was significantly down-regulated following fluvoxamine augmentation. Additionally, the clinical assessments showed improvement in negative symptoms following the combined treatment. These findings suggested that gene expression changes in PMC's may be useful in investigating the mechanism of drug action in schizophrenia.

In this study we will examine RNA and protein expression in the course of fluvoxamine augmentation treatment. 15 chronic schizophrenic patients who have persistent negative symptoms and cognitive impairment despite adequate treatment will participate. Fluvoxamine 100mg/day will be added to the treatment regimen and continued for 6 weeks. Clinical state will be assessed using validated rating scales and cognitive performance will be assessed with a cognitive test battery. Blood samples will be taken at baseline and at 1, 3 and 6 weeks. The PMC's will be assayed using microarray, RT PCR and proteomic techniques. Changes in RNA and protein expression will be detected and compared with changes in clinical symptoms and cognitive function. Identification of biochemical changes related to augmentation treated and their relation to symptomatic and cognitive changes will be the major potential benefit of the study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* A diagnosis of schizophrenia (DSM-IVTR)
* Antipsychotic dose unchanged for at least 2 weeks prior to study
* SANS score>= 3 on at least one of the global measures of affective blunting, alogia or avolition.
* Knowledge of Hebrew

Exclusion Criteria:

* Dementia or other serious neurological disorders
* History of alcohol or drug use
* Patients with a legal guardian
* Patients involuntarily hospitalized by order of the district psychiatrist
* Use of antidepressants within 1 month of the study
* Renal or hepatic disorder
* Patients with upper GI bleeds
* Patients with SIADH syndrome
* Pregnant woman

Criteria for the cessation of the study after initial commencement:

* Severe adverse events (including but not only GI, cardiovascular, neurologic, hematologic or urologic severe adverse events)
* Emergent suicidality
* Emergence of hypomanic or manic symptoms
* If the subject requests to stop

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2008-04; Primary Completion 2009-04 (Estimated); Study Completion 2009-04 (Estimated)

PRIMARY OUTCOMES:
Schedule for the Assessment of Negative Symptoms (SANS) | 0 weeks, 3 weeks, 6 weeks

SECONDARY OUTCOMES:
Schedule for the Assessment of Positive Symptoms (SAPS) | 0 weeks, 3 weeks, 6 weeks
Simpson Angus Scale for Extrapyramidal Side Effects (SA) | 0 weeks, 3 weeks, 6 weeks
Abnormal Involuntary Movement Scales (AIMS) | 0 weeks, 3 weeks, 6 weeks
Calgary Depression Scale | 0 weeks, 3 weeks, 6 weeks
Mini Mental State Examination | 0 weeks, 3 weeks, 6 weeks
Dot test (Keefe et al., 1997) | 0 weeks, 3 weeks, 6 weeks
Digit Span (Wechsler, 1998) | 0 weeks, 3 weeks, 6 weeks
Finger Tap Test (Reitan and Davison, 1974) | 0 weeks, 3 weeks, 6 weeks
Wechsler memory tests (Wechsler, 1998) | 0 weeks, 3 weeks, 6 weeks
Computerized Cognitive Neuropsychological Battery (Silver et al 2003) | 0 weeks, 3 weeks, 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Henry Silver, PhD, Principal Investigator — Sha'ar Menshae Mental Health Center
Locations (1):
- Sha'ar Menashe Mental Health Center, Mobile Post Hefer, Israel

REFERENCES:
- [Background] Ackenheil M. The mechanism of action of antidepressants revised. J Neural Transm Suppl. 1990;32:29-37. doi: 10.1007/978-3-7091-9113-2_3. PMID 2089097
- [Background] Addington D, Addington J, Schissel B. A depression rating scale for schizophrenics. Schizophr Res. 1990 Jul-Aug;3(4):247-51. doi: 10.1016/0920-9964(90)90005-r. PMID 2278986
- [Background] Andreasen NC. The Scale for the Assessment of Negative Symptoms (SANS): conceptual and theoretical foundations. Br J Psychiatry Suppl. 1989 Nov;(7):49-58. No abstract available. PMID 2695141
- [Background] Avissar S, Roitman G, Schreiber G. Differential effects of the antipsychotics haloperidol and clozapine on G protein measures in mononuclear leukocytes of patients with schizophrenia. Cell Mol Neurobiol. 2001 Dec;21(6):799-811. doi: 10.1023/a:1015164423918. PMID 12043849
- [Background] Chalifour LE, Fahmy R, Holder EL, Hutchinson EW, Osterland CK, Schipper HM, Wang E. A method for analysis of gene expression patterns. Anal Biochem. 1994 Feb 1;216(2):299-304. doi: 10.1006/abio.1994.1045. PMID 7513971
- [Background] Chertkow Y, Weinreb O, Youdim MB, Silver H. The effect of chronic co-administration of fluvoxamine and haloperidol compared to clozapine on the GABA system in the rat frontal cortex. Int J Neuropsychopharmacol. 2006 Jun;9(3):287-96. doi: 10.1017/S1461145705005626. Epub 2005 Jun 21. PMID 15967061
- [Background] Chertkow Y, Weinreb O, Youdim MB, Silver H. Dopamine and serotonin metabolism in response to chronic administration of fluvoxamine and haloperidol combined treatment. J Neural Transm (Vienna). 2007;114(11):1443-54. doi: 10.1007/s00702-007-0753-1. Epub 2007 Jun 18. PMID 17576515
- [Background] Chertkow Y, Weinreb O, Youdim MB, Silver H. Gene expression changes in peripheral mononuclear cells from schizophrenic patients treated with a combination of antipsychotic with fluvoxamine. Prog Neuropsychopharmacol Biol Psychiatry. 2007 Oct 1;31(7):1356-62. doi: 10.1016/j.pnpbp.2007.04.016. Epub 2007 Apr 29. PMID 17662512
- [Background] Debouck C, Goodfellow PN. DNA microarrays in drug discovery and development. Nat Genet. 1999 Jan;21(1 Suppl):48-50. doi: 10.1038/4475. PMID 9915501
- [Background] de Saizieu A, Certa U, Warrington J, Gray C, Keck W, Mous J. Bacterial transcript imaging by hybridization of total RNA to oligonucleotide arrays. Nat Biotechnol. 1998 Jan;16(1):45-8. doi: 10.1038/nbt0198-45. PMID 9447592
- [Background] DeRisi JL, Iyer VR, Brown PO. Exploring the metabolic and genetic control of gene expression on a genomic scale. Science. 1997 Oct 24;278(5338):680-6. doi: 10.1126/science.278.5338.680. PMID 9381177
- [Background] Duman RS, Malberg J, Thome J. Neural plasticity to stress and antidepressant treatment. Biol Psychiatry. 1999 Nov 1;46(9):1181-91. doi: 10.1016/s0006-3223(99)00177-8. PMID 10560024
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Goff DC, Midha KK, Sarid-Segal O, Hubbard JW, Amico E. A placebo-controlled trial of fluoxetine added to neuroleptic in patients with schizophrenia. Psychopharmacology (Berl). 1995 Feb;117(4):417-23. doi: 10.1007/BF02246213. PMID 7604142
- [Background] Guy W (ed). National Institute of Mental Health. Abnormal Involuntary Movement Scale (AIMS). Early Clinical Drug Evaluation Unit Assessment Manual. Rockville, Maryland: US Department of Health and Human Services, 1976; pp. 534-537
- [Background] Ilani T, Ben-Shachar D, Strous RD, Mazor M, Sheinkman A, Kotler M, Fuchs S. A peripheral marker for schizophrenia: Increased levels of D3 dopamine receptor mRNA in blood lymphocytes. Proc Natl Acad Sci U S A. 2001 Jan 16;98(2):625-8. doi: 10.1073/pnas.98.2.625. Epub 2001 Jan 9. PMID 11149951
- [Background] Keefe RS, Lees-Roitman SE, Dupre RL. Performance of patients with schizophrenia on a pen and paper visuospatial working memory task with short delay. Schizophr Res. 1997 Jul 25;26(1):9-14. doi: 10.1016/S0920-9964(97)00037-6. PMID 9376341
- [Background] Kronfol Z, Remick DG. Cytokines and the brain: implications for clinical psychiatry. Am J Psychiatry. 2000 May;157(5):683-94. doi: 10.1176/appi.ajp.157.5.683. PMID 10784457
- [Background] Lesch KP, Aulakh CS, Wolozin BL, Tolliver TJ, Hill JL, Murphy DL. Regional brain expression of serotonin transporter mRNA and its regulation by reuptake inhibiting antidepressants. Brain Res Mol Brain Res. 1993 Jan;17(1-2):31-5. doi: 10.1016/0169-328x(93)90069-2. PMID 8381906
- [Background] Lesch KP, Manji HK. Signal-transducing G proteins and antidepressant drugs: evidence for modulation of alpha subunit gene expression in rat brain. Biol Psychiatry. 1992 Oct 1;32(7):549-79. doi: 10.1016/0006-3223(92)90070-g. PMID 1333286
- [Background] Peiffer A, Veilleux S, Barden N. Antidepressant and other centrally acting drugs regulate glucocorticoid receptor messenger RNA levels in rat brain. Psychoneuroendocrinology. 1991;16(6):505-15. doi: 10.1016/0306-4530(91)90034-q. PMID 1811246
- [Background] Pepin MC, Pothier F, Barden N. Antidepressant drug action in a transgenic mouse model of the endocrine changes seen in depression. Mol Pharmacol. 1992 Dec;42(6):991-5. PMID 1480137
- [Background] Reitan RM, Davison LA. Clinical Neuropsychology: Current Status and Applications. New York, New York: 1974, Hemisphere
- [Background] Andreasen NC. Scale for the Assessment of Positive Symptoms (SAPS). 1983, Iowa City. The University of Iowa
- [Background] Rothermundt M, Arolt V, Bayer TA. Review of immunological and immunopathological findings in schizophrenia. Brain Behav Immun. 2001 Dec;15(4):319-39. doi: 10.1006/brbi.2001.0648. PMID 11782102
- [Background] Silver H, Nassar A. Fluvoxamine improves negative symptoms in treated chronic schizophrenia: an add-on double-blind, placebo-controlled study. Biol Psychiatry. 1992 Apr 1;31(7):698-704. doi: 10.1016/0006-3223(92)90279-9. No abstract available. PMID 1599987
- [Background] Silver H, Shmugliakov N. Augmentation with fluvoxamine but not maprotiline improves negative symptoms in treated schizophrenia: evidence for a specific serotonergic effect from a double-blind study. J Clin Psychopharmacol. 1998 Jun;18(3):208-11. doi: 10.1097/00004714-199806000-00005. PMID 9617979
- [Background] Silver H, Feldman P, Bilker W, Gur RC. Working memory deficit as a core neuropsychological dysfunction in schizophrenia. Am J Psychiatry. 2003 Oct;160(10):1809-16. doi: 10.1176/appi.ajp.160.10.1809. PMID 14514495
- [Background] Simpson GM, Angus JW. A rating scale for extrapyramidal side effects. Acta Psychiatr Scand Suppl. 1970;212:11-9. doi: 10.1111/j.1600-0447.1970.tb02066.x. No abstract available. PMID 4917967
- [Background] Spina E, De Domenico P, Ruello C, Longobardo N, Gitto C, Ancione M, Di Rosa AE, Caputi AP. Adjunctive fluoxetine in the treatment of negative symptoms in chronic schizophrenic patients. Int Clin Psychopharmacol. 1994 Winter;9(4):281-5. doi: 10.1097/00004850-199400940-00007. PMID 7868850
- [Background] Toth M, Shenk T. Antagonist-mediated down-regulation of 5-hydroxytryptamine type 2 receptor gene expression: modulation of transcription. Mol Pharmacol. 1994 Jun;45(6):1095-100. PMID 7517496
- [Background] Wechsler D. Wechsler Adult Intelligence Scale Manual. New York, New York: Guilford Press, 1998; pp. 95-188